CLINICAL TRIAL: NCT02691143
Title: The Effect of TheraBand® Kinesiology Tape on Post-manipulation Pain and Range of Motion
Acronym: TBKTManip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSR07
Record Dates: First submitted 2016-02-15; First posted 2016-02-25 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-01

CONDITIONS: Acute Non-complicated Postural Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manipulation plus Tape (Experimental): The Tape Group will have TheraBand® Kinesiology Tape, an elastic therapeutic tape (ETT), applied immediately following cervical manipulation from a licensed chiropractor. The taping protocol will be applied by the investigator and consist of a "Y" strip applied at 25% tension running superior to inferior from the hair line to T1-2 and a horizontal "I" strip applied at 50% tension at the site of pain.
  Interventions: Other: TheraBand Kinesiology Tape
- Manipulation Only (No Intervention): The control group will receive manipulation from a licensed chiropractor only

INTERVENTIONS:
Other: TheraBand Kinesiology Tape — One approach to treating musculoskeletal conditions is a elastic therapeutic taping technique designed to target muscles and lymphatic system. Limited research on the efficacy of elastic therapeutic taping (ETT) is available for specific patient populations, including neck pain. ETT it is theorized to impact muscle function by inhibiting or facilitating the muscle, improve blood flow, reduce pain, and improve joint alignment. In a study by Gonzalez-Iglesias et al. the investigators reported that neck pain and range of motion significantly improved immediately and 24 hours after the application of ETT in acute whiplash patients as compared to a sham taping.
  Arms: Manipulation plus Tape

SUMMARY:
The purpose of this study is to determine if post-manipulation elastic therapeutic tape (ETT) with TheraBand® Kinesiology Tape to neck pain patients can impact neck range of motion (ROM) and post-manipulation pain. A convenience sample of 50 patients, between the ages of 18-64, who present with acute non-complicated postural neck pain will be recruited from an outpatient chiropractic clinic. Upon providing consent to participate, patients will be randomly assigned into 2 groups; Control Group (manipulation only) and Tape Group (manipulation plus tape). Pain and neck ROM will be recorded at 3 different intervals: (1) pre-cervical manipulation, (2) within 5 minutes of cervical manipulation, (3) with 24-48 hours after manipulation.

DETAILED DESCRIPTION:
The purpose of this study is to determine if post-manipulation elastic therapeutic tape (ETT) with TheraBand® Kinesiology Tape to neck pain patients can impact neck range of motion (ROM) and post-manipulation pain. A convenience sample of 50 patients, between the ages of 18-64, who present with acute non-complicated postural neck pain will be recruited from an outpatient chiropractic clinic. Complications would include discogenic pain or radicular symptoms. Inclusionary criteria would also consist of onset less than 18 days and the indications for cervical manipulation, including pain, decreased range of motion, and hypertonicity. Exclusionary criteria will include pregnancy, contraindications to manipulation, and previous neck surgery. Patients will be recruited on the first visits to ensure they haven't receive manipulation before for this current plan of care. Upon providing consent to participate, patients will be randomly assigned into 2 groups; Control Group (n=25) and Tape Group (n=25). Pain and neck ROM will be recorded at 3 different intervals: (1) pre-cervical manipulation, (2) within 5 minutes of cervical manipulation, (3) with 24-48 hours after manipulation. The control group will receive manipulation only, while the Tape Group will have ETT TheraBand® Kinesiology Tape applied immediately following cervical manipulation. The taping protocol will be applied by the investigator and consist of a "Y" strip applied at 25% tension running superior to inferior from the hair line to T1-2 and a horizontal "I" strip applied at 50% tension at the site of pain. Six cervical ranges of motion values will be recorded utilizing the Acumar DataCapture hand-held dual inclinometer. Range of motion will be measured at maximum (max) degrees and average degrees of 6 trials and will include: flexion (F), extension €, left side-bending (LSB), right side-bending (RSB), left rotation (LR), and right rotation (RR). Measure of pain will be asked of each patient using the Numeric Pain Rating Scale (NPRS) from 0-10. They will be asked to rate their pain at rest and when in motion.

ELIGIBILITY:
Inclusion criteria will include ages of 18-64 who present with non-complicated postural neck pain, indications for cervical manipulation, including pain, decreased range of motion, and hypertonicity. Exclusion criteria will include discogenic pain or radicular symptoms, pregnancy, contraindications to manipulation, and previous neck surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jena Slaski, MEd, ATC, Study Director — Sport and Spine Rehab Clinical Research Foundation
Locations (1):
- Sport and Spine Rehab, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A convenience sample of who presented with acute non-complicated neck pain were recruited from an outpatient chiropractic clinic
Groups:
- Manipulation Plus Tape: The Tape Group had TheraBand® Kinesiology Tape, an elastic therapeutic tape (ETT), applied immediately following cervical manipulation from a licensed chiropractor. The taping protocol was applied by the investigator and consist of a "Y" strip applied at 25% tension running superior to inferior from the hair line to T1-2 and a horizontal "I" strip applied at 50% tension at the site of pain.
- Manipulation Only: The control group received manipulation from a licensed chiropractor only
Period: Overall Study
Arm/Group | Manipulation Plus Tape | Manipulation Only
Started | 27 | 23
Completed | 27 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manipulation Plus Tape | Manipulation Only | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Continuous [Mean (Full Range); unit: years] | 36.9 [20 to 61] | 36.5 [18 to 58] | 36.7 [20 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Cervical Range of Motion
Description: Six cervical ranges of motion values will be recorded utilizing the Acumar DataCapture hand-held dual inclinometer. Range of motion will be measured at maximum (max) degrees and average degrees of 6 trials and will include: flexion (F), extension (E), left side-bending (LSB), right side-bending (RSB), left rotation (LR), and right rotation (RR).
Time Frame: 3 Testing sessions: (T1) Baseline, (T2) Immediate Post, and (T3) 24-48hours
Measure: Mean (Full Range); unit: degrees
Arm/Group | Manipulation Plus Tape | Manipulation Only
Number analyzed (Participants) | 27 | 23
degrees
  T1 Flexion Max | 37.9 [5 to 64] | 36.9 [12 to 50]
  T2 Flexion Max | 39.5 [17 to 58] | 37.5 [17 to 50]
  T3 Flexion Max | 42.44 [19 to 55] | 39 [9 to 62]
  T1 Extension Max | 34.3 [17 to 45] | 32.4 [11 to 46]
  T2 Extension Max | 36.5 [17 to 51] | 38.7 [22 to 65]
  T3 Extension Max | 41.7 [15 to 60] | 36.9 [16 to 52]
  T1 Left Side Bending Max | 27.9 [4 to 49] | 28 [15 to 43]
  T2 Left Side Bending Max | 30.5 [1 to 45] | 33.7 [8 to 61]
  T3 Left Side Bending Max | 36.7 [12 to 62] | 32.2 [16 to 50]
  T1 Right Side Bending Max | 31.6 [10 to 49] | 32.7 [19 to 53]
  T2 Right Side Bending Max | 35.3 [21 to 54] | 34.5 [15 to 60]
  T3 Right Side Bending Max | 39 [21 to 62] | 35.1 [14 to 58]
  T1 Left Rotation Max | 54.5 [22 to 99] | 51.7 [24 to 87]
  T2 Left Rotation Max | 53.2 [18 to 86] | 53.2 [17 to 83]
  T3 Left Rotation Max | 52.8 [27 to 86] | 50 [22 to 94]
  T1 Right Rotation Max | 52.6 [17 to 78] | 50.2 [20 to 85]
  T2 Right Rotation Max | 53.8 [16 to 72] | 50.9 [20 to 90]
  T3 Right Rotation Max | 56.5 [15 to 78] | 52.5 [14 to 93]

2. Secondary Outcome: Change in Numeric Pain Rating Scale (NPRS)
Description: Subjects rate their pain on the Numeric Pain Rating Scale (NPRS), a scale from 0-10, 0 being none and 10 being the worst imaginable.
Time Frame: 3 Testing sessions: (T1) Baseline, (T2) Immediate Post, and (T3) 24-48hours
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Manipulation Plus Tape | Manipulation Only
Number analyzed (Participants) | 27 | 23
units on a scale
  T1 Pain | 6.1 [2 to 9] | 5.7 [2 to 9]
  T2 Pain | 5.4 [2 to 8] | 5 [2 to 9]
  T3 Pain | 4.9 [1 to 8] | 4.9 [1 to 9]

ADVERSE EVENTS:
Arm/Group | Manipulation Plus Tape | Manipulation Only
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/23
Other Adverse Events (participants affected / at risk) | 0/27 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes